CLINICAL TRIAL: NCT03674138
Title: Pharmacogenomic-Guided Antidepressant Drug Prescribing in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-19578
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Depression; Anxiety; Generalized Anxiety Disorder; Depressive Disorder; Major Depressive Disorder; Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Generalized Anxiety Disorder; Depressive Disorder; Depressive Disorder, Major; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to the genomic results for 12 weeks, with the 12 week time period starting at the time of antidepressant drug prescribing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DNA-guided choice of therapy (Active Comparator): DNA-guided choice of antidepressant therapy
  Interventions: Diagnostic Test: DNA-guided choice of therapy
- Clinical management (Active Comparator): Clinical management
  Interventions: Diagnostic Test: DNA-guided choice of therapy; Other: Clinical management

INTERVENTIONS:
Diagnostic Test: DNA-guided choice of therapy — Buccal swab for DNA genotyping to identify best antidepressant therapy
Other: Clinical management — Clinical management to identify best antidepressant therapy
  Arms: Clinical management

SUMMARY:
This is a prospective, randomized clinical trial to investigate the clinical impact of a preemptive pharmacogenomics strategy to guide antidepressant therapy in cancer patients. Those enrolled onto the clinical trial will be randomized to either DNA-guided choice of therapy or clinical management alone. Scores on self-reported measures of depressive and anxiety symptoms along with quality of life will be compared between cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cancer diagnosis
* Be 18 years of age or older
* Patients who rate depression or anxiety > 5 based on a 10 point scale
* Patients expected to live greater than 6 months
* Serum bilirubin and creatinine < 1.5x upper limit of normal
* AST and ALT < 3 times upper limit of normal
* Willing and able to provide written informed consent
* Able to complete self-assessment questionnaires

Exclusion Criteria:

* Patients not diagnosed with cancer
* Antidepressant prescribing performed by a non-Moffitt psychiatrist after enrollment onto the clinical trial
* Known Pregnancy
* History of liver or allogenic stem cell transplant
* Patients with a known cognitive impairment (e.g., delirium, dementia, etc.) or psychological impairment (e.g., schizophrenia, bipolar disease, etc.) other than depressive and anxiety symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms from baseline, as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, week 12, month 12
  The Hospital Anxiety and Depression scale can range from 0 to 42 (14 questions each on a 0-3 point scale).
Change in anxious symptoms from baseline, as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, week 12, month 12
  The Hospital Anxiety and Depression scale can range from 0 to 42 (14 questions each on a 0-3 point scale).

SECONDARY OUTCOMES:
Quality of Life as measured by Functional Assessment of Cancer Therapy-General (FACT-G) Scale | 12 months
  Quality of Life as measured by Functional Assessment of Cancer Therapy-General (FACT-G) Scale. FACT-G is a quality of life questionnaire with values ranging from 0 (not at all) to 4 (very much). The categories of measure are physical, social/family, emotional and functional well-being.

CONTACTS AND LOCATIONS:
Overall Officials: James K Hicks, PharmD, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States